CLINICAL TRIAL: NCT02494063
Title: A Prospective Observational Trial on Sentinel Lymph Node Biopsy in Patients With Early Stage Cervical Cancer
Brief Title: Sentinel Lymph Node Biopsy in Patients With Early Stages Cervical Cancer
Acronym: SENTIX
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, David Cibula, MD, PhD, Professor, Charles University, Czech Republic
Other Study IDs: CEEGOG CX-01; ENGOT-Cx 2 (Other: ENGOT); CEEGOG CX-01 (Other: Central and Eastern European Gynecologic Oncology Group); Protocol v2.0 (1st amendment) (Other: EC approval (VI.2018)); Protocol v3.0 (2nd amendment) (Other: EC approval (XII.2020)); Protocol v3.1 (3rd amendment) (Other: EC approval (VII.2021)); 16-31643A (Other Grant/Funding Number: Czech Research Council); 19-03-00023 (Other Grant/Funding Number: Czech Research Council)
Record Dates: First submitted 2015-07-06; First posted 2015-07-10 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; sentinel lymph node; lymphadenectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sentinel lymph node (SLN): Only sentinel lymph node biopsy, no further pelvic lymph nodes removal, radical hysterectomy.
  Interventions: Procedure: Sentinel lymph node biopsy
- Control: Control group is composed by either those who were enrolled into the trial, but who did not fulfil intra-operative criteria (especially failure to detect SLN on both pelvic side walls) or those in whom systematic lymphadenectomy is planned upfront.
  Interventions: Procedure: At least unilateral systematic pelvic lymph node dissection

INTERVENTIONS:
Procedure: Sentinel lymph node biopsy — Bilateral sentinel lymph node biopsy, pathologic ultrastaging
  Groups: Sentinel lymph node (SLN)
Procedure: At least unilateral systematic pelvic lymph node dissection
  Groups: Control

SUMMARY:
To evaluate whether a less radical surgical approach with sentinel lymph node biopsy is non-inferior to treatment with systematic pelvic lymphadenectomy.

The null hypothesis is that the recurrence rate after SLN biopsy is non-inferior to the reference recurrence rate of 7 % (at the 24th month of follow-up) in patients after systematic pelvic lymphadenectomy, but that the less radical surgery is associated with significantly lower postoperative morbidity.

DETAILED DESCRIPTION:
Patients will be enrolled in the study at the time of surgery planning; at this point, a patient´s consent will be requested if inclusion criteria are fulfilled (histological type, FIGO stage, age, performance status, lymph node clinical status). The following procedures will be provided prior to surgery: clinical staging (MRI or EUS), medical data collection, adverse events assessment, lymphedema assessment, quality of life questionnaire, ECOG performance status, weight and height, standard pre-operative laboratory workup, pregnancy test if clinically indicated.

Surgery should be done within 6 weeks of the imaging study (MRI or expert US). During the surgery, local or distant cancer spread outside of the cervix will be excluded, SLN will be detected, and all SLN will be sent for intra-operative pathologic evaluation. In patients with SLN detection on both sides of the pelvis no other lymph nodes will be removed and they will continue in the study. SLN biopsy will be followed by radical hysterectomy (type B, C1, or C2) or fertility-sparing procedure, according to the pre-operative plan.

Intra-operatively, three groups of patient will be excluded from the SLN study group (though they can be included in the control group):

1. Patients with intra-operative detection of more advanced disease stage (> IB1)
2. Patients with failure to detect SLN bilaterally (either no SLN detected or only on one side of the pelvis)
3. Patients with intra-operative pathologic detection of macrometastases or micrometastases in SLN

In these patients who were excluded from the study group, further surgery and adjuvant treatment will be provided according to the institutional guidelines. These patients will remain in a database and reasons for their exclusion from the SLN study group will be entered into the SIS (Form 2).

A control group will be established to compare postoperative morbidity in patients after SLN biopsy only and after complete pelvic lymphadenectomy. Patients in whom complete lymphadenectomy was performed at least on one side of the pelvis will be eligible for the control group.

In patients, who continue in the study, all SLNs will be processed by pathologists according to the protocol for SLN ultrastaging (Chapter 7.4.2; Appendix 11). If macrometastases or micrometastases or isolated tumor cells are detected in any of the SLNs by pathologic ultrastaging after the surgery, adjuvant radiotherapy will be recommended to the patient. No adjuvant treatment will be offered to those with negative final lymph node status, confirmed pre-operative disease FIGO stage (IA1 - IB1), and adequately performed radical hysterectomy with negative parametrial and vaginal margins.

Follow-up will consist of visits at regular intervals of 6 months after the surgery (additional visits in shorter intervals can be scheduled according to institutional guidelines). The following procedures will be provided at each visit during the follow-up period: pelvic examination, symptomatic lymphocele assessment, quality of life assessment (6 and 12 months after the surgery), adverse events assessment, and secondary lower extremity lymphedema assessment (maximum 6 years after surgery in SLN group, 4 years in Control group). Other imaging studies will be done only if clinically indicated. Any postoperative complication or disease recurrence will be managed according to the institutional guidelines.

Outcomes after fertility sparing procedures in selected centres with be collected (i.e. morbidity after cervical procedure or ovarian transposition, treatment of infertility, pregnancy rates and complications).

ELIGIBILITY:
I) SLN study group:

Inclusion criteria:

A) Preoperative:

1. FIGO stage IA1+LVSI; IA2; IB1
2. No evidence of bulky or suspicious pelvic lymph nodes or distant metastases in preoperative conventional imaging studies
3. Performance status ECOG: 0 - 1
4. Age ≥ 18 years, ≤ 75 years
5. Squamous cell carcinoma OR Adenocarcinoma usual type (HPV related)
6. Suitable candidates for primary surgical treatment such as:

   * radical hysterectomy in tumors ≤ 4 cm in the largest diameter OR
   * fertility-sparing treatment in tumors ≤ 2 cm in the largest diameter
7. History of second primary cancer only if > 5 years with no evidence of disease
8. Approved and signed Informed consent

B) Intra-operative

1. Bilateral SLN detection
2. Negative intra-operative pathologic SLN evaluation (frozen section)
3. No intra-operative evidence of more advanced disease (>IB1)

Exclusion Criteria:

1. Neoadjuvant chemotherapy
2. Pregnancy
3. History of pelvic or abdominal radiotherapy
4. HIV positivity / AIDS
5. Adenosquamous cancer or adenocarcinoma unusual type (non HPV related - such as: mucinous, clear cell, mesonephric)

II) Control Group:

Inclusion criteria:

A) Preoperative:

1. FIGO stage IA1 + LVSI; IA2; IB
2. Performance status ECOG: 0-1
3. Age ≥ 18 years, ≤ 75 years
4. Patient is not pregnant
5. No history of pelvic or abdominal radiotherapy
6. Patient scheduled for surgical treatment including systematic pelvic lymphadenectomy
7. Approved and signed Informed Consent

B) Intra-operative:

a) Systematic pelvic lymphadenectomy performed at least on one side of the pelvis

Exclusion criteria:

1. Pregnancy
2. History of pelvic or abdominal radiotherapy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early stages cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-06; Primary Completion 2022-12 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
Recurrence rate at the 24th month of follow-up (cervical recurrences after fertility-sparing procedures will be excluded) | 24 months
  Recurrence rate (RR) will be estimated at the 24th month of follow-up to prove a non-inferiority of SLN biopsy to the reference value (RR 24th month: 7 %).

SECONDARY OUTCOMES:
Prevalence of symptomatic pelvic lymphocele | 2 years
  Reduction in the prevalence of at least 30% to the reference prevalence (6%).
Prevalence of lower extremity lymphedema | 2 years
  Reduction in the prevalence of at least 30% to the reference prevalence (30%).
Postoperative morbidity | 2 years
  Early postoperative morbidity (30 days after surgery) will be evaluated using 5-grade "Dindo" Classification of surgical complications. Late postoperative morbidity (from 30 days up to 2 years after surgery) will be evaluated using Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
DFS (Disease-free survival) | 2 years
  Disease-free survival after treatment with primary surgery until first recurrence.
Pelvic DFS (Pelvic Disease-free survival) | 2 years
  Disease-free survival after treatment with primary surgery until first recurrence within the pelvis.
Quality of life (QoL) | 1 year
  The quality of life (QoL) will be assessed by European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 self-administered multi-dimensional scale cancer specific questionnaire, which is validated in 81 languages. It consists of 5 function scales, three symptom scales, six single-items and a global QoL score.
Intra-operative morbidity | 1 month
  Intra-operative morbidity will be evaluated using 5-grade "Dindo" Classification of surgical complications.
FNR (False Negative Rate) of intra-operative pathologic SLN evaluation | 2 years
  Proportion of patients with lymph nodes negative on intraoperative evaluation but positive on final ultrastaging
DFS in SLN negative patients | 2 years
  Disease free survival in patients with SLN negative on final ultrastaging
Recurrence rate safety margins | 2 years
  Recurrence rate safety margin (> 0.12) as the study stopping rule will be examined when the first 30, 60,150 and 300 patients complete the 12-month follow-up.
Overall survival | 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: David Cibula, MD, Principal Investigator — Gynecologic Oncology Center, Department of Obstetrics and Gynecology, General University Hospital and 1st Faculty of Medicine, Charles University Prague, Czechia
Locations (1):
- Gynecologic Oncology Center in Prague, Prague, Czechia

REFERENCES:
- [Background] Zikan M, Fischerova D, Pinkavova I, Slama J, Weinberger V, Dusek L, Cibula D. A prospective study examining the incidence of asymptomatic and symptomatic lymphoceles following lymphadenectomy in patients with gynecological cancer. Gynecol Oncol. 2015 May;137(2):291-8. doi: 10.1016/j.ygyno.2015.02.016. Epub 2015 Feb 24. PMID 25720294
- [Background] Cibula D, Oonk MH, Abu-Rustum NR. Sentinel lymph node biopsy in the management of gynecologic cancer. Curr Opin Obstet Gynecol. 2015 Feb;27(1):66-72. doi: 10.1097/GCO.0000000000000133. PMID 25502426
- [Background] Giammarile F, Bozkurt MF, Cibula D, Pahisa J, Oyen WJ, Paredes P, Olmos RV, Sicart SV. The EANM clinical and technical guidelines for lymphoscintigraphy and sentinel node localization in gynaecological cancers. Eur J Nucl Med Mol Imaging. 2014 Jul;41(7):1463-77. doi: 10.1007/s00259-014-2732-8. Epub 2014 Mar 8. PMID 24609929
- [Background] Cibula D, Abu-Rustum NR, Dusek L, Slama J, Zikan M, Zaal A, Sevcik L, Kenter G, Querleu D, Jach R, Bats AS, Dyduch G, Graf P, Klat J, Meijer CJ, Mery E, Verheijen R, Zweemer RP. Bilateral ultrastaging of sentinel lymph node in cervical cancer: Lowering the false-negative rate and improving the detection of micrometastasis. Gynecol Oncol. 2012 Dec;127(3):462-6. doi: 10.1016/j.ygyno.2012.08.035. Epub 2012 Aug 31. PMID 22943880
- [Background] Cibula D, Abu-Rustum NR, Dusek L, Zikan M, Zaal A, Sevcik L, Kenter GG, Querleu D, Jach R, Bats AS, Dyduch G, Graf P, Klat J, Lacheta J, Meijer CJ, Mery E, Verheijen R, Zweemer RP. Prognostic significance of low volume sentinel lymph node disease in early-stage cervical cancer. Gynecol Oncol. 2012 Mar;124(3):496-501. doi: 10.1016/j.ygyno.2011.11.037. Epub 2011 Nov 25. PMID 22120175
- [Background] Cibula D, Abu-Rustum NR, Benedetti-Panici P, Kohler C, Raspagliesi F, Querleu D, Morrow CP. New classification system of radical hysterectomy: emphasis on a three-dimensional anatomic template for parametrial resection. Gynecol Oncol. 2011 Aug;122(2):264-8. doi: 10.1016/j.ygyno.2011.04.029. Epub 2011 May 17. PMID 21592548
- [Background] Cibula D, Abu-Rustum NR. Pelvic lymphadenectomy in cervical cancer--surgical anatomy and proposal for a new classification system. Gynecol Oncol. 2010 Jan;116(1):33-7. doi: 10.1016/j.ygyno.2009.09.003. Epub 2009 Oct 17. PMID 19837449
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Derived] Cibula D, Marnitz S, Jarkovsky J, Kocian R, Dundr P, Klat J, Zapardiel I, Arencibia O, Landoni F, Presl J, Raspagliesi F, Zikan M, van Lonkhuijzen LR, Torne A, Slama J, Minar L, Ostojich M, Pilka R, Petiz AF, Petzel A, Burgetova A, Fischerova D, Nemejcova K, Kohler C. Sentinel lymph node biopsy without systematic pelvic lymphadenectomy in females with early-stage cervical cancer: final outcome of the SENTIX prospective, single-arm, noninferiority, international trial. Nat Cancer. 2025 Sep;6(9):1585-1594. doi: 10.1038/s43018-025-01016-y. Epub 2025 Jul 4. PMID 40615729
- [Derived] Borcinova M, Kohler C, Nemejcova K, Zapardiel I, Klat J, Fruhauf F, Kalist V, Szatkowski W, Wydra D, Kocian R, Laky R, Toth R, Misiek M, Redecha M, Martin I, Kridelka F, Burgetova A, Santiago Garcia FJ, Van Gorp T, Szewczyk G, Kipp B, Poka R, Coronado PJ, Cadron I, Luyckx M, Fischerova D, Fischbach R, Cibula D. Preoperative tumour size assessment in patients with early-stage cervical cancer: Final results of the SENTIX study. Gynecol Oncol. 2025 May;196:160-167. doi: 10.1016/j.ygyno.2025.04.005. Epub 2025 Apr 11. PMID 40220456
- [Derived] Cibula D, Kohler C, Jarkovsky J, Kocian R, Dundr P, Klat J, Zapardiel I, Landoni F, Fruhauf F, Fischbach R, Borcinova M, Fischerova D. Magnetic resonance imaging and ultrasound examination in preoperative pelvic staging of early-stage cervical cancer: post-hoc analysis of SENTIX study. Ultrasound Obstet Gynecol. 2025 Apr;65(4):495-502. doi: 10.1002/uog.29205. Epub 2025 Mar 25. PMID 40130299
- [Derived] Kocian R, Kohler C, Bajsova S, Jarkovsky J, Zapardiel I, Di Martino G, van Lonkhuijzen L, Sehnal B, Sanchez OA, Gil-Ibanez B, Martinelli F, Presl J, Minar L, Pilka R, Kascak P, Havelka P, Michal M, van Gorp T, Nemejcova K, Dundr P, Cibula D. Sentinel lymph node pathological ultrastaging: Final outcome of the Sentix prospective international study in patients with early-stage cervical cancer. Gynecol Oncol. 2024 Sep;188:83-89. doi: 10.1016/j.ygyno.2024.06.015. Epub 2024 Jun 27. PMID 38941963
- [Derived] Borcinova M, Ragosch V, Jarkovsky J, Bajsova S, Pilka R, Glickman A, Garrido-Mallach S, Raspagliesi F, Szatkowski W, Pakiz M, Snyman LC, Kocian R, Tamussino K, Kalist V, Michal M, Segovia MG, Poka R, Kipp B, Szewczyk G, Wydra D, Toth R, Vinnytska A, Fischerova D, Siegler K, Cibula D. Challenges in lower limb lymphoedema assessment based on limb volume change: Lessons learnt from the SENTIX prospective multicentre study. Gynecol Oncol. 2022 Jan;164(1):76-84. doi: 10.1016/j.ygyno.2021.10.089. Epub 2021 Nov 8. PMID 34763939
- [Derived] Cibula D, Kocian R, Plaikner A, Jarkovsky J, Klat J, Zapardiel I, Pilka R, Torne A, Sehnal B, Ostojich M, Petiz A, Sanchez OA, Presl J, Buda A, Raspagliesi F, Kascak P, van Lonkhuijzen L, Barahona M, Minar L, Blecharz P, Pakiz M, Wydra D, Snyman LC, Zalewski K, Zorrero C, Havelka P, Redecha M, Vinnytska A, Vergote I, Tingulstad S, Michal M, Kipp B, Slama J, Marnitz S, Bajsova S, Hernandez A, Fischerova D, Nemejcova K, Kohler C. Sentinel lymph node mapping and intraoperative assessment in a prospective, international, multicentre, observational trial of patients with cervical cancer: The SENTIX trial. Eur J Cancer. 2020 Sep;137:69-80. doi: 10.1016/j.ejca.2020.06.034. Epub 2020 Aug 1. PMID 32750501
- [Derived] Cibula D, Dusek J, Jarkovsky J, Dundr P, Querleu D, van der Zee A, Kucukmetin A, Kocian R. A prospective multicenter trial on sentinel lymph node biopsy in patients with early-stage cervical cancer (SENTIX). Int J Gynecol Cancer. 2019 Jan;29(1):212-215. doi: 10.1136/ijgc-2018-000010. PMID 30640706